CLINICAL TRIAL: NCT00429832
Title: A Randomized Controlled Trial of Ondansetron and Promethazine in the Treatment of Nausea and Vomiting in the Emergency Department
Brief Title: A RCT of Ondansetron and Promethazine in the Treatment of Nausea and Vomiting in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-006
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: Nausea; Vomiting
Keywords: Nausea, vomiting, antiemetic
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron; Promethazine

INTERVENTIONS:
Drug: Ondansetron
Drug: promethazine

SUMMARY:
This was a trial comparing two commonly used medications for nausea and vomiting, ondansetron and promethazine, in the Emergency Department.

DETAILED DESCRIPTION:
Nausea and vomiting are common complaints in the emergency department (ED). There are many pharmacologic agents used for the treatment of these complaints. None are new nor experimental. Very little research has been done in the ED setting to determine which of these agents is most effective with the least adverse effects. Our own previous research found that droperidol but not prochlorperazine and metoclopramide is more effective than placebo. Because of the recent FDA black box warning added to droperidol, the use of this agent has suddenly ceased in many EDs. Promethazine remains a very commonly used antiemetic in many EDs but one recent study found it less effective than prochlorperazine which was in turn found no more effective than placebo in our own study. As a result many physicians have turned to ondansetron, a newer and more expensive agent. Experience among anesthesiologists and oncologists has shown ondansetron to be highly effective with a minimum of adverse effects. These patient populations, however, are very different from those found in the ED. It is our hypothesis that promethazine and ondansetron are equally effective for the ED treatment of unselected patients with nausea and vomiting with similar rates of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Chief complaint of nausea or vomiting

Exclusion Criteria:

* Age less than 18
* unable to provide informed consent
* rate nausea at < 40 mm on 100 mm VAS
* received antiemetic within 24 hours
* pregnant or possibly pregnant
* reported allergy to either study medication
* received more than 1 liter of intravenous fluids
* their primary ED physician declined to have patient participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-10; Study Completion 2005-11

PRIMARY OUTCOMES:
Reduction in nausea on a VAS.

SECONDARY OUTCOMES:
Change in sedation on a VAS
Change in anxiety on a VAS
Need for rescue medication at 30 minutes
Patient satisfaction at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Darren A Braude, MD, MPH, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital Emergency Department, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Braude D, Crandall C. Ondansetron versus promethazine to treat acute undifferentiated nausea in the emergency department: a randomized, double-blind, noninferiority trial. Acad Emerg Med. 2008 Mar;15(3):209-15. doi: 10.1111/j.1553-2712.2008.00060.x. PMID 18304050